CLINICAL TRIAL: NCT04587908
Title: A Phase 3, Randomized, Placebo-controlled, Double-blind and Open-label, Extension Study of TAS-205 in Patients With Duchenne Muscular Dystrophy
Brief Title: A Phase 3 Study of TAS-205 in Patients With Duchenne Muscular Dystrophy（REACH-DMD）
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10053050
Record Dates: First submitted 2020-10-13; First posted 2020-10-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — TAS-205; Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAS-205 (Experimental)
  Interventions: Drug: TAS-205 [Ambulatory Cohort] [Non-ambulatory Cohort]
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo [Ambulatory Cohort] only

INTERVENTIONS:
Drug: TAS-205 [Ambulatory Cohort] [Non-ambulatory Cohort] — ・Treatment period：oral administration for 52 weeks, BID after meal
  Arms: TAS-205
Drug: Placebo [Ambulatory Cohort] only — * Observation period：oral administration for 2 weeks, BID after meal
  * Treatment period：oral administration for 52 weeks, BID after meal
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TAS-205 in patients with Duchenne muscular dystrophy

DETAILED DESCRIPTION:
[Ambulatory Cohort] The main purpose of this cohort is to assess the efficacy of TAS-205 in patients with Duchenne muscular dystrophy (DMD) compared with placebo as measured by the mean change from baseline to 52 weeks in the time to rise from the floor． Following completion of the treatment period, patients may elect to continue in open-label extension study.

[Non-ambulatory Cohort] The main purpose of this cohort is to assess the safety of TAS-205 in patients with DMD by collecting the incidence of adverse events for 52 weeks.

ELIGIBILITY:
Key Inclusion Criteria [Ambulatory Cohort]

* Patients with a diagnosis of dystrophinopathy as determined by a dystrophin genetic test at the time of informed consent, symptoms or signs characteristic to DMD (e.g., proximal muscular weakness, waddling gait, Gower's sign)
* Patients aged 5 years or more at the time of informed consent
* Patients weighing more than 7.5 kg and less than 60 kg at the time of screening test
* Patients who meet all of the following at the time of screening test
* walk by themselves
* time to rise from the floor on own is ≥ 3 seconds and <10 seconds
* Patients who can expect a 6-minute walking test of 350 meters or more
* If taking oral glucocorticoids no significant change in the total daily or dosing 6 months before enrollment.

[Non-ambulatory Cohort]

* Patients with a diagnosis of DMD as determined by a dystrophin genetic test at the time of informed consent.
* Patients weighing more than 7.5 kg and less than 90 kg at the time of screening test
* Patients who meet all of the following criteria as definition of non-ambulatory at the time of enrollment
* Use of a wheelchair on a daily basis.
* No orthopedic pathology (fracture, sprain, injury, etc.) or acute deterioration associated with surgical treatment.
* Inability to walk 10 meters within 30 seconds on the 10-meter run/walk test at enrollment.
* Patients with a Brooke Score of 5 or less in the arm and shoulder at enrollment.
* Patients who are able to take the drug orally throughout the treatment period (crushed or suspended doses are not acceptable)
* If taking oral glucocorticoids no significant change in the total daily or dosing 90 days prior to obtaining consent, or not taking oral glucocorticoids for more than 90 days prior to obtaining consent and whose symptoms are stable.
* Patients on angiotensin-converting enzyme inhibitors, beta-blockers, and angiotensin II receptor blockers for the treatment (including prophylaxis) of heart failure who are symptomatically stable with no change in dosage (prescription basis) within 90 days prior to enrollment.

Key exclusion Criteria [Ambulatory Cohort]

* Patients who have serious concomitant drug hypersensitivity or medical history
* Patients who have used cyclooxygenase-1 (COX-1) or COX-2 inhibitors, or nonsteroidal anti-inflammatory drugs (NSAIDs) during 7 days before the measurement of time to rise from the floor in the screening period
* Patients who have incurred an injury (trauma/damage) that may affect muscle strength or motor function within 3 months before enrollment or who have an uncured injury (trauma/damage) that may affect muscle strength or motor function at the enrollment
* Patients who have received gene-/cell-based therapy or stop-codon readthrough therapy with antisense oligonucleotides
* Patients who have participated in another clinical trial and received a study drug within 90 days before study drug administration in the present study
* Patients with a left ventricular ejection fraction (EF) of <40% or left ventricular fractional shortening (FS) of <25% on the cardiac ultrasonography (echocardiography) at observation period

[Non-ambulatory Cohort]

* Patients with severe cardiac disease (including a history of pacemaker surgery)
* Patients with left ventricular EF <40% on echocardiography within 14 days prior to enrollment
* Patients with %FVC less than 40% within 14 days prior to enrollment
* Patients with respiratory diseases such as asthma, bronchitis, COPD, bronchiectasis, emphysema, pneumonia, etc. (including chronic use of beta2 agonists, inhaled steroids, sympathomimetics, anticholinergic agents, etc.)
* Patients on continuous ventilator use (excluding use while sleeping)
* Patients who have undergone surgery within 180 days prior to enrollment that may affect muscle strength or exercise, pulmonary function, or cardiac function, or are planning such surgery during the study period
* Injury (trauma/injury) within 90 days prior to enrollment that may affect muscle strength or motor, pulmonary, or cardiac function, or that has not healed at the time of enrollment
* Patients who are judged by the principal investigator or subinvestigator to have brain dysfunction such as intellectual disability, autistic tendencies, and attention deficit hyperactivity disorder that would interfere with the performance of efficacy and safety evaluation
* Patients with systemic allergic or chronic inflammatory diseases that may interfere with the interpretation of efficacy or safety data (except allergic rhinitis, localized or mild atopic dermatitis, eczema, etc.)
* Patients enrolled in Treatment Phase Part A of this study's Ambulatory Cohort

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline to Week 52 in the time to rise from the floor | Baseline to Week 52 of treatment
  Ambulatory Cohort
Incidence of Adverse Events and Adverse Reactions | Week 52
  Non-ambulatory Cohort

SECONDARY OUTCOMES:
Time measured in the time to rise from the floor test, as well as the change from baseline in each measured value | Baseline to 52 weeks of treatment
  Ambulatory Cohort
Change from baseline in the Timed Up and Go Test (TUG) | Baseline to 52 weeks of treatment
  Ambulatory Cohort Timed Up and Go Test (TUG) The time required for the subject to stand up from a sitting position on a table (chair), walk to a cone placed 3 m ahead as quickly as possible, and then return to the table will be evaluated.
  The time required for the subject to stand up from a sitting position on a table (chair), walk to a cone placed 3 m ahead as quickly as possible, and then return to the table will be evaluated.
Change from baseline in North Star Ambulatory Assessment (NSAA) | Baseline to 52 weeks of treatment
  Ambulatory Cohort
Change from baseline in Six-minutes Walk Test (6MWT) | Baseline to 52 weeks of treatment
  Ambulatory Cohort
Measured values of Muscle volume index (MVI), Percent Muscle volume index (%MVI) and skeletal muscle mass in skeletal muscle computed tomography (CT), as well as the change from baseline in each measured value | Baseline to 52 weeks of treatment
  Ambulatory Cohort
Assessment of upper limb function: The Brooke upper extremity scale, measured values of performance of the upper limb (PUL) and change from baseline in measured values | week 52
  Non-ambulatory Cohort
Change from baseline in grip strength | week 52
  Non-ambulatory Cohort
Pulmonary function tests: measured effort lung capacity (FVC, %FVC), volume in 1 second (Forced Expiratory Volume :FEV1.0), fraction in 1 second (FEV1.0%), and change from baseline (at enrollment) of measured values. | week 52
  Non-ambulatory Cohort
Echocardiography: Measured EF and FS and change from baseline in measured values | week 52
  Non-ambulatory Cohort

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (5):
- Japan (5):
  - A site selected by Taiho Pharmaceutical Co., Ltd., Aichi
  - A site selected by Taiho Pharmaceutical Co., Ltd., Fukuoka
  - A site selected by Taiho Pharmaceutical Co., Ltd., Hokkaido
  - A site selected by Taiho Pharmaceutical Co., Ltd., Osaka
  - A site selected by Taiho Pharmaceutical Co., Ltd., Tokyo

IPD SHARING:
Plan to Share IPD: No
Data will not be shared according to the Sponsor policy on data sharing. Taiho policy on data sharing may be found at https://www.taiho.co.jp/en/science/policy/clinical_trial_information_disclosure_policy/index.html.